CLINICAL TRIAL: NCT06210191
Title: Intramedullary Headless Screw Fixation for Metacarpal and Phalangeal Fractures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelrahman Megahed Ahmed, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Intramedullary screw fixation
Record Dates: First submitted 2023-12-18; First posted 2024-01-18 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Metacarpal Fracture; Phalanx Fracture
Keywords: intramedullary headless screw fixation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- union of fracture (Experimental): Intramedullary headless screw fixation for metacarpal and phalangeal fractures
  Interventions: Procedure: Intramedullary headless screw fixation

INTERVENTIONS:
Procedure: Intramedullary headless screw fixation — fixation of fractures of metacarpals and phalanges by intramedullary headless screws

SUMMARY:
Intramedullary headless screw fixation for metacarpal and phalangeal fractures

DETAILED DESCRIPTION:
The most frequent fractures in the upper extremities are phalangeal and metacarpal fractures accounts about 40%, which follow distal radius fractures in order of frequency.

There are many methods of fixation of these fractures as plates and K-wires. Plate fixation is able to provide open reduction and stability for early range of motion with mixed clinical results. Reported complications include stiffness, fixed flexion contracture of the adjacent joints, soft tissue dissection, and extensor lag.

There are minimally invasive techniques, including the use of K-wires, lag screws, cerclage wiring, and external fixation that limit soft tissue dissection. These options have drawbacks of malunion, nonunion, infection, need for hardware removal, and stiffness.

Intramedullary headless screw fixation is an emerging alternative to K-wire or plate fixation of displaced and unstable fractures of the phalanges and metacarpals. The Intramedullary headless screw fixation is a new option that offers rigid stability, early active range of motion, and easy insertion. Due to the minimally invasive nature of this technique, patients will experience better results in terms of range of motion, return to work faster, and minimize complications.

Beck et al. reported 100% of patients achieved full radiological union with minor complication rate and full range of motion and early return to work with average 96% of grip strength.

ELIGIBILITY:
Inclusion Criteria:

1. Skeletally mature patients with closed fractures of phalanges and metacarpals.
2. Patients with open type I fractures of phalanges and metacarpals.

Exclusion Criteria:

1. Skeletally immature patients with open physis.
2. Patients with open type II or III fractures of phalanges or metacarpals.
3. Patients with fractures of phalanges or metacarpals with neurovascular injury. 4 Patients with associated tendon injuries.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Achieve full range of motion of hand joints | 6 weeks for active range of motion
  Change DASH Score of hand functions to 0 by this intervention. As 0 is excellent and 100 is the worst outcome

CONTACTS AND LOCATIONS:
Overall Officials: Amr Elsayed, professor, Study Chair — Assiut University; Waleed Riad, professor, Study Director — Assiut University
Locations (1):
- Faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available. all collected IPD, all IPD that underlie results in a publication)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting in January 2025 or as a date relative to the time when summary data are published
Access Criteria: access criteria of my IPD will be available with my investigators